CLINICAL TRIAL: NCT06259981
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, and Tolerability of GLY-200 in Participants With Obesity
Brief Title: A 16-Week Study to Evaluate the Efficacy, Safety, and Tolerability of GLY-200 in Participants With Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glyscend, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GLY-200-03
Record Dates: First submitted 2024-01-31; First posted 2024-02-14 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Obesity
Keywords: Obesity; Glyscend, Inc.; GLY-200
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GLY-200 (Experimental): Participants will receive 2.0 g GLY-200 orally twice daily for 16 weeks.
  Interventions: Drug: GLY-200
- Placebo (Placebo Comparator): Participants will receive placebo (identical in appearance to GLY-200) orally twice daily for 16 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLY-200 — 2.0 g GLY-200 (4 x 0.5 g capsules) orally twice daily
  Arms: GLY-200
Drug: Placebo — 4 placebo capsules orally twice daily
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy, safety, and tolerability of GLY-200 in participants with obesity.

DETAILED DESCRIPTION:
This study is a Phase 2, randomized, double-blind, placebo-controlled, multi-center study in adult participants with obesity. Approximately 70 participants will be randomized in a 1:1 ratio to GLY-200 (2.0 g, twice daily) or placebo (twice daily). There will be a ≤ 28-day screening period. Dosing will occur for 16 weeks. Clinic visits will occur at Screening, Week 0 (Day 1), and Weeks 1, 2, 4, 6, 8, 12, 16, and 17 [End of Study (EOS)] or Early Termination (ET). Phone visits will occur at Week 3, 10, and 14.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ≥ 18 and ≤ 70 years old at the time of screening
* BMI ≥ 32 and ≤ 40 kg/m² at screening

Exclusion Criteria:

* Known history of any form of diabetes mellitus, or HbA1c ≥6.5% (48 mmol/mol)
* Participants who have had an increase or decrease in body weight more than 5% within the last 3 months
* Treated with any prescription medication or procedure that promotes weight loss or weight gain in the last 6 months
* Use of any drug treatment that affects gastric pH
* Use of any drug treatment that affects gastrointestinal motility
* Diagnosis or treatment of any symptomatic or structural abnormality of the GI tract or active disease within 12 months
* Clinically significant symptoms (as determined by the Investigator) of nausea, vomiting, bloating, diarrhea, flatulence, constipation, or abdominal pain in the last 30 days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2024-10-23 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in weight | Baseline and Week 16
Proportion of participants who achieve ≥ 5% body weight reduction | Baseline and Week 16

SECONDARY OUTCOMES:
Change and percent change from baseline in weight | Baseline, Week 1, Week 2, Week 4, Week 6, Week 8, Week 12, and Week 16
Change from baseline in waist circumference | Baseline, Week 1, Week 2, Week 4, Week 6, Week 8, Week 12, and Week 16
Incidence of adverse events (AEs) and serious adverse events (SAEs) considered by the Investigator to be related to study drug administration | Over the 16-week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Mark Fineman, PhD, Study Chair — Glyscend, Inc.
Locations (5):
- United States (5):
  - Tampa Bay Medical Research, Inc., Clearwater, Florida
  - Sensible Healthcare, LLC, Ocoee, Florida
  - Tandem Clinical Research, Marrero, Louisiana
  - Mercury Street Medical, Butte, Montana
  - Clinical Trials of Texas, Inc., San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No